CLINICAL TRIAL: NCT01080040
Title: Observational Study to Assess the Prevalence of Spasticity and the Impact on the Quality of Life in Patients With Multiple Sclerosis in Argentina
Brief Title: To Assess the Prevalence of Spasticity and the Impact on the Quality of Life in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200077-507
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis, Relapsing Remitting
Keywords: Multiple Sclerosis, Relapsing Remitting; Quality of life
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is observational, non-controlled, multicentric and prospective, without experimental intervention or control. As part of the usual management of the subjects, scales will be used for the assessment of the spasticity and the quality of life (QoL).

The purpose of this observational study is to assess the incidence of spasticity in a group of subjects with Relapsing Remitting Multiple Sclerosis (RRMS) in Argentina and the way it affects the QoL of these subjects.

DETAILED DESCRIPTION:
One of most frequently observed symptoms in subjects with MS is spasticity. Spasticity is defined as an abnormal velocity-dependent increase in muscle tonic stretch reflexes due to an amplified reactivity of motor segments to sensory input. It is part of one of the components of the superior motoneurone syndrome and it may cause muscle rigidity and disability.

The spasticity, which could be measured in electrophysiological, biomechanical and clinical terms, has a significant prevalence. It is a frequent cause for consultation among subjects with MS and, consequently, has a significant impact on the QoL. Men and those subjects with MS of longer duration are the most affected by spasticity.

The aim of this study is to assess the impact that spasticity has on the QoL of subjects with MS.

The total duration of the study is 24 months. The recruiting period will be 12 months. Once the recruiting time is over, the collection of data will continue during the full 24 months period that was planned.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 21 60 years of age
* Subjects with established diagnosis of RRMS according to the revised McDonald criteria - 2005
* Subjects with a diagnosis of RRMS for more than one year
* The subject who have signed the Informed Consent

Exclusion Criteria:

* Subjects with other causes of spasticity
* Subjects with other clinical forms of MS (different from relapsing-remitting)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with established diagnosis of RRSM for more than one year.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assess the prevalence of spasticity in subjects with RRMS | Initial visit (Day 0) to 24 months
  Ashworth Scale (AS) (Spasticity) Expanded Disability status scale (EDSS) SF 36

SECONDARY OUTCOMES:
Evaluation of the impact of spasticity on the quality of life of subjects with RRMS | Initial visit (Day 0) to 24 months
Evaluation of the changes in spasticity after 24 months | Initial visit (Day 0) to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jose A. Brizuela, Principal Investigator — Fundación Rosarina de Neurorehabilitación. Rosario, Argentina.
Locations (1):
- Fundación Rosarina de Neurorehabilitación, Rosario, Argentina